CLINICAL TRIAL: NCT02098512
Title: A Multicenter Pilot Study of Reduced Intensity Conditioning and Allogeneic Stem Cell Transplantation Followed by Targeted Immunotherapy in Children, Adolescents and Young Adults With Poor Risk CD30+ Hodgkin Lymphoma (HL)
Brief Title: Immunotherapy Following Reduced Intensity Conditioning and Allogeneic Stem Cell Transplant for Poor Risk CD30+ Hodgkin Lymphoma Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Medical College (Other)
Collaborators: St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 564
Record Dates: First submitted 2014-03-17; First posted 2014-03-28 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Hodgkin Lymphoma
Keywords: Brentuximab Vedotin; Immunotherapy; Relapsed Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Reduced Intensity Conditioning; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Transplant and Immunotherapy (Experimental): We intend to utilize reduced intensity conditioning and allogeneic stem cell transplant from HLA matched sibling or unrelated adult donor followed by post-AlloSCT Brentuximab Vedotin in patients with poor risk Hodgkin Lymphoma.
  Interventions: Drug: Brentuximab Vedotin; Procedure: Allogeneic Stem Cell Transplantation; Drug: Reduced Intensity Conditioning

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin will be administered every 21 days starting on or around Day +42 post allogeneic stem cell transplant for a TOTAL of 4 doses as outlined below:
  * 42 (+/-7 days) Brentuximab Vedotin 1.8 mg/kg (max=180 mg) IV x 1
  * 63 (+/- 7 days) Brentuximab Vedotin 1.8 mg/kg (max=180 mg) IV x 1
  * 84 (+/- 7 days) Brentuximab Vedotin 1.8 mg/kg (max = 180 mg) IV x 1
  * 105 (+/- 7 days) Brentuximab Vedotin 1.8 mg/kg (max=180 mg) IV x 1
  Other Names: Adcetris
Procedure: Allogeneic Stem Cell Transplantation — Following conditioning with chemotherapy, patients will receive stem cells from a matched related or unrelated donor.
Drug: Reduced Intensity Conditioning — Patients will receive reduced intensity chemotherapy with one of three regimens: Busulfan/Fludarabine; Gemcitabine/Fludarabine/Melphalan; Fludarabine/Cyclophosphamide

SUMMARY:
Patients with relapsed or refractory Hodgkin Lymphoma who are CD30+ will receive a standard of care reduced intensity regimen and an allogeneic stem cell transplant (from another person, related or unrelated). Following recovery, patients will receive a medication called Brentuximab Vendotin which is targeted against CD30+ cells. The study hypothesis is that this treatment will be safe and well tolerated in children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or less.
* Patients with Hodgkin Lymphoma with either of the following:

  • Primary induction failure (failure to achieve initial CR) and/or primary refractory disease OR First, Second or Third relapse AND History of prior ablative auto HSCT or ineligible for an ablative auto HSCT or ≥25% residual disease after at least two reinduction chemotherapy cycles AND HLA matched family donor (6/6 or 5/6) or matched unrelated adult donor (MUD) (8/8) or matched umbilical cord blood unit (≥5/6) with prethaw cell dose of at least 3 x 107/kg TNC.
* off other investigational therapy for one month prior to entry in this study.
* adequate organ function

Exclusion Criteria:

* Patients with HD with 4th or greater CR, PR, and/or SD are ineligible.
* Patients with rapidly progressive disease (PD) unresponsive to reinduction chemo, radio, or immunotherapy are ineligible.
* Patients who don't have an eligible donor are ineligible.
* Women who are pregnant are ineligible.

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 1 year
  Patients will be followed for one year for adverse events related to the administration of study drug.
Overall Survival | 1 year
  patients will be assessed for one year to determine survival status

SECONDARY OUTCOMES:
To assess feasibility of developing a bank of LMP-specific CTLs from healthy donors | 3 years
  A bank of from identified EBV positive donors will be established for potential use in current and future clinical trials in LMP-positive lymphomas. Annual review will occur to assess the feasibility of recruiting healthy donors to help build this cell line bank. If there are no cell lines developed within the first year, an alternative design may be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States